CLINICAL TRIAL: NCT02005939
Title: Effect of Pomegranate Extract Intake on Anthropometric, Metabolic and Hormonal Parameters in Human Volunteers: a Double Blinded, Placebo Controlled, Randomised, Exploratory 4 Week Trial.
Brief Title: Effect of Biophenol-rich Pomegranate Extract Intake on Blood Pressure, Hormones, Body Composition and Quality of Life in Healthy Volunteers.
Acronym: POM-01Expl
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Margaret University (Other)
Collaborators: PomeGreat (Unknown)
Responsible Party: Principal Investigator, Angela Stockton, P.h.D. Researcher, Queen Margaret University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: POM-01Expl; POM-01Expl (Other: Queen Margaret University)
Record Dates: First submitted 2013-12-04; First posted 2013-12-09 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Cardiovascular Risk Factors
Keywords: Pomegranate; Blood pressure; Insulin sensitivity; Cortisol; Quality of life; Body composition
MeSH Terms: conditions — Insulin Resistance | interventions — pomegranate fruit rind

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pomegranate extract capsule (Experimental): All participants receive 1.1 g pomegranate extract capsule daily for 4 weeks
  Interventions: Dietary Supplement: Pomegranate extract
- Placebo capsule (Placebo Comparator): All participants receive a 1.1g placebo capsule daily for 4 weeks

INTERVENTIONS:
Dietary Supplement: Pomegranate extract — All randomised participants to the intervention arm receive one pomegranate capsule daily for 4 weeks
  Other Names: Pomegreat PurePlus
  Arms: Pomegranate extract capsule

SUMMARY:
Biophenols can act as powerful antioxidants. Pomegranate (Punica granatum) provides a rich and varied source of biophenols with the most abundant being ellagitannins, tannins, anthocyanins, ellagic and gallic acids. Interest in antioxidant polyphenol-rich pomegranate products has increased in recent years with growing reports of potential health benefits. Pomegranate biophenols have been noted to lower systolic blood pressure, salivary stress hormones and increase insulin sensitivity in previous trials involving participants who have cardiovascular disease, but few studies have been conducted recruiting healthy volunteers, and those have made use of pomegranate juice rather than extract.

The aim of this parallel study is to investigate the effect of pomegranate extract supplementation on blood pressure, lipid profiles, salivary stress hormones, insulin sensitivity, body composition and the perceived quality of life in healthy volunteers over 4 weeks.

It hypothesizes that consumption of biophenol-rich Pomegranate extract could increase insulin sensitivity and perceived quality of life while decreasing blood pressure, body measurements and stress hormones in healthy individuals.

DETAILED DESCRIPTION:
After randomisation to a study arm, eligible participants will consume either one pomegranate extract or placebo capsule (identical in appearance) daily, for a period of 4 weeks. The pomegranate capsule contains 650mg of pomegranate extract (240 mg punicalagins and 350mg total biophenols) and the placebo, maltodextrin.

Participants will be required to attend the university clinic lab twice, having fasted overnight, with all measurements being taken pre and post study at 4 weeks. Blood, saliva and 24 hr urine samples will be provided. Body weight and composition, dietary habits and quality of life will also be measured. The well validated health related Quality of Life Questionnaire (Rand 36) will be administered pre- and post-intervention. This series of questions covers eight spheres of health. The physical health component considers physical functioning, physical role, bodily pain and general health. The mental health aspect examines vitality, social functioning, emotional role and general mental health. Anthropometric measurements recorded will be height, weight, waist, mid upper arm circumference. Bioelectrical impedance analysis (BIA), which measures conductivity from hand to foot, calculating both body fat and fat free mass, will also be performed.

Pre and post study comparison of the amount of polyphenols in 24 hr urine samples provided, alongside capsule consumption checks, will measure compliance. A 3 day diet diary record, will be used for recording energy intake and to highlight any fluctuations in dietary intake over the study period.

The data will be analysed using Statistical Programme for Social Sciences (SPSS) for Windows software version 19. Differences in baseline characteristics will be examined using independent t- tests with extract and placebo groups as independent variables and outcome measures as dependent variables. Paired t-tests will determine any individual differences between pre and post biochemical markers and anthropometric measurements. ANCOVAs will determine the overall differences between the independent groups.

This exploratory study will provide a foundation for and refine the outcome measures required for a larger future trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants
* BMI from 18-35
* Males and Females
* Age: 18-65 years

Exclusion Criteria:

Systemic disease, including heart disease and diabetes

* Allergic reactions
* Alcohol/drug abuse
* Immunological conditions
* Pregnancy or lactation
* Liver and kidney disease
* Management for weight control within the last 2 months
* Heavy smokers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Blood pressure | Week 0, 4
  Change in systolic and diastolic blood pressure

SECONDARY OUTCOMES:
Changes in insulin sensitivity | Week 0, 4
  Measured through fasting insulin and glucose

OTHER OUTCOMES:
stress hormone levels | Week 0, 4
  Measured via saliva using ELISA methods
Changes in body composition | week 0, 4
  Assessed via BMI, body fat mass
Quality of Life | Week 0, 4
  Assessed by the scored Rand 36 Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Emad AS Al-Dujaili, Ph.D., Study Director — Queen Margaret University
Locations (1):
- Queen Margaret University, Edinburgh, Scotland, United Kingdom